CLINICAL TRIAL: NCT05512533
Title: Feasibility and Safety of Thin Convex Probe EBUS Scope BF-UC290F for the Diagnosis of Peripheral Pulmonary Lesions
Brief Title: Feasibility of Thin Cp-EBUS Scope BF-UC290F for the Diagnosis of PPLs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Jiayuan Sun, Director, Department of Endoscopy, Shanghai Chest Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SHCHE202208
Record Dates: First submitted 2022-08-21; First posted 2022-08-23 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Peripheral Pulmonary Lesions
Keywords: EBUS-TBNA; diagnostic yield; peripheral pulmonary lesions (PPLs)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BF-UC290F for diagnosing PPLs (Experimental): Thin EBUS endoscope is inserted and used to visualize peripheral pulmonary lesions, and biopsies will be conducted by EBUS-TBNA.
  Interventions: Device: Linear Ultrasound Bronchoscope BF-UC290F (Olympus)

INTERVENTIONS:
Device: Linear Ultrasound Bronchoscope BF-UC290F (Olympus) — A thin Olympus EBUS bronchoscope BF-UC290F will be used for all endobronchial ultrasound examinations, and biopsies will be conducted with EBUS needles - the ViziShot 2 22G (Olympus).

SUMMARY:
The purpose of the study is to evaluate the diagnostic value and safety of Thin Convex Probe Endobronchial Ultrasound (TCP-EBUS) Scope for peripheral pulmonary lesions (PPLs)

DETAILED DESCRIPTION:
This study will determine the feasibility of the novel thin convex probe endobronchial ultrasound (TCP-EBUS) Scope for the diagnosis of peripheral pulmonary lesions. The primary end point is to clarify the feasibility of using the thin convex probe EBUS scope to biopsy peripheral pulmonary lesions. The secondary objective is to evaluate operation time, sample adequacy, factors affecting the diagnosis rate, etc. The safety, insertion ability, and operability of the thin convex probe EBUS would also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years old.
* Chest imaging shows the presence of peripheral pulmonary lesions (surrounded by pulmonary parenchyma and located below the segmental bronchus as seen radiographically.) suspicious of malignancy, 0.8-5cm in greatest diameter in need of bronchoscopic biopsy for clinical purposes, and the investigators consider it possible to be biopsied with BF-UC290F (the bronchus adjacent or leading to the PPLs are close to 5mm in diameter, thus BF-UC290F is able to arrival/access).
* Patients without contraindications of bronchoscopy.
* Patients have good medical adherence and signed informed consent.

Exclusion Criteria:

* Peripheral pulmonary lesion is pure ground-glass opacity.
* Visible lumen lesions during bronchoscopy
* The lesions were adjacent to the central airway (trachea, left and right main bronchus, and right middle bronchus), and the biopsies by the Thin Convex Probe EBUS Scope BF-UC290F were conducted without leaf bronchus entry
* The investigators believe that patient has other conditions that are not suitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-09-02 (Actual); Primary Completion 2023-02-12 (Actual); Study Completion 2023-07-12 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield of BF-UC290F for PPLs | Up to 6 months
  Diagnostic yield is defined as the proportion of peripheral pulmonary lesions (PPLs) diagnosed via endobronchial ultrasound-guided transbronchial needle aspiration (EBUS-TBNA) in all lesions undergoing bronchoscopy biopsy via EBUS-TBNA.

SECONDARY OUTCOMES:
EBUS scope operation time | Immediately after each operation
  It is defined as the total time from insertion of the EBUS scope to withdrawal of the EBUS scope
The total time of lesion access | Immediately after Each Operation
  It is defined as the total time from the insertion of the EBUS scope to the arrival confirmed by ultrasound image.
Factors affecting the diagnosis rate | Up to 6 months
  Factors affecting the diagnosis rate, including the nature of the lesions, the size of the lesions, the location of the lesions and so on will be analyzed.
The bronchus level of lesions, and the bronchus level reached with the EBUS scope | During the procedure
  Level: Main bronchus is level 0, lobar bronchus is level 1, segment bronchus is level 2, sub-segment bronchus is level 3, and so on, such as: LB3a is level 3
Specimen adequacy | Up to 6 months
  The adequacy of specimens obtained by Thin Convex Probe EBUS Scope BF-UC290F for pathological typing, molecular testing, and immune checkpoint detection

OTHER OUTCOMES:
Safety Outcome: Complication rate | 1 month
  The complications refer to the total of serious adverse events related to the procedure during or within 1 month after the operation

CONTACTS AND LOCATIONS:
Overall Officials: Jiayuan Sun, MD., PhD., Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhi X, Wang L, Chen J, Zheng X, Li Y, Sun J. Scoring model of convex probe endobronchial ultrasound multimodal imaging in differentiating benign and malignant lung lesions. J Thorac Dis. 2020 Dec;12(12):7645-7655. doi: 10.21037/jtd-2020-abpd-005. PMID 33447457
- [Background] Fujino K, Ujiie H, Kinoshita T, Lee CY, Igai H, Inage T, Motooka Y, Gregor A, Suzuki M, Yasufuku K. First Evaluation of the Next-Generation Endobronchial Ultrasound System in Preclinical Models. Ann Thorac Surg. 2019 May;107(5):1464-1471. doi: 10.1016/j.athoracsur.2018.11.068. Epub 2019 Jan 2. PMID 30610852